CLINICAL TRIAL: NCT04139044
Title: The Effects of Unilateral Balance Training on Bilateral Balance and Explosive Power Among Athletes With Chronic Ankle Instability
Brief Title: The Effects of Unilateral Balance Training Among Athletes With Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YeditepeUptr
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Ankle Injuries; Ankle Sprains
Keywords: ankle, joint instability, cross-education, rehabilitation
MeSH Terms: conditions — Ankle Injuries; Joint Instability

STUDY DESIGN:
Intervention Model Description: The sample of the study consists of athletes with a history of CAI who registered as a team player at Yeditepe University Culture and Sports Directorate between February 2019 and June 2019.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stable Ankle Training Group (SG) (Experimental): Balance Exercise Training for Only The Stable Ankle
  Interventions: Procedure: Balance Exercise Training for Stable Ankle
- Unstable Ankle Training Group (UG) (Experimental): Balance Exercise Training for Only The Unstable Ankle
  Interventions: Procedure: Balance Exercise Training for Unstable Ankle
- Control Group (CG) (No Intervention): No balance exercise training

INTERVENTIONS:
Procedure: Balance Exercise Training for Stable Ankle — Balance and hop stabilization exercises were administered for 30 minutes of each exercise session.
  Arms: Stable Ankle Training Group (SG)
Procedure: Balance Exercise Training for Unstable Ankle — Balance and hop stabilization exercises were administered for 30 minutes of each exercise session.
  Arms: Unstable Ankle Training Group (UG)

SUMMARY:
The aim of the study is to investigate the effects of a 4-week, unilateral balance exercise training program on bilateral balance and explosive power in athletes with chronic ankle instability. The participants were randomly divided into Stable Ankle Training Group (SG) (n=9), Unstable Ankle Training Group (UG) (n=9) and control group (CG) (n=10). The balance exercise training program was administered for only the stable ankle of athletes in SG and only the unstable ankle of athletes in UG, twice a week and for a 4-week duration.

DETAILED DESCRIPTION:
The aim of the study is to investigate the effects of a 4-week, unilateral balance exercise training program on bilateral balance and explosive power in athletes with chronic ankle instability (CAI). The study included 28 volunteer athletes with a history of CAI who registered as a team player at Yeditepe University Culture and Sports Directorate February 2019 - June 2019. The severity of functional ankle instability of all the athletes was assessed by the Cumberland Ankle Instability Tool (CAIT). Functional limitations of the athletes with CAI were evaluated by Foot and Ankle Ability Measure Activity of Daily Living Subscale (FAAM-ADL) and Sports Subscale (FAAM-S). Balance Error Scoring System (BESS) was used to determine the static balance performance of athletes. Dynamic balance was evaluated by the Y Balance Test (YBT). Sport performance including vertical jumping and hopping was assessed with Single-Legged Countermovement Jump (CMJ) Test, Figure-of-Eight Hop Test, and Side Hop Test. The athletes were randomly divided into Rehabilitation for the Stable Ankle Group (SG) (n=9), Rehabilitation for the Unstable Ankle Group (UG) (n=9) and Control Group (CG) (n=10). Athletes in SG and UG were included balance exercise training program. The balance exercise training program was administered for only the stable ankle of athletes in SG and only the unstable ankle of athletes in UG, twice a week and for a 4-week duration.

ELIGIBILITY:
Inclusion Criteria:

* Participating in the study on a voluntary basis
* Athletes with 18-25 years old
* Being a player in one of the basketball, volleyball, and handball team sports
* Athletes with a history of at least 2 significant lateral ankle sprains which were classified as a second degree and related to inflammatory symptoms (pain, swelling)
* The self-reported sensation of giving away and instability at the injured ankle confirmed by the Cumberland Ankle Instability Tool with a score ≤25
* Recurrent lateral ankle sprain episodes of the injured ankle occurred at least 12 months
* The self-reported function of the injured ankle confirmed by Foot and Ankle Ability Measure with a score <90% from activities of daily living subscale and <80% from sport subscale.

Exclusion Criteria:

* A history of surgery to the musculoskeletal structures in either lower extremity
* A history of a fracture in either lower extremity necessitating realignment
* Acute injury of musculoskeletal structures of other joints of the lower extremity in the previous 3 months affecting joint function and integrity
* Presence of bilateral ankle instability
* Balance or vestibular disorder

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Foot and Ankle Ability Measure | 4 weeks
  The FAAM is a self-reported tool improved to evaluate the physical functions of individuals with musculoskeletal disorders related to foot and ankle.
Balance Error Scoring System | 4 weeks
  The BESS is a valid test to find out deficits in static postural control of individuals with CAI.
Y Balance Test | 4 weeks
  The Y Balance Test is the functional test that is able to find out impairments in dynamic postural control among individuals with CAI
Single-Leg Countermovement Jump Test | 4 weeks
  The Single-LegCountermovement jump test is used to evaluate the lower-extremity power of athletes, and indirectly the functional performance.
Figure-of-Eight Hop Test | 4 weeks
  Figure-of-8 Hop Test is used to measure the explosive power of the lower extremity of athletes.
Side Hop Test | 4 weeks
  Side Hop test is a test used to evaluate the explosive power of the lower extremity of athletes.

SECONDARY OUTCOMES:
Cumberland Ankle Instability Tool | Baseline
  Cumberland Ankle Instability Tool including a 30-point scale of 9-items is a valid and reliable questionnaire for distinguishing and quantifying the severity of functional instability.

CONTACTS AND LOCATIONS:
Overall Officials: Ayça Yağcıoğlu, MSc, Principal Investigator — Yeditepe University, Health Sciences Faculty, Physiotherapy and Rehabilitation; Gökhan Metin, Professor, Study Chair — Istanbul University, Faculty of Medicine, Sports Medicine; Feryal Subaşı, Professor, Study Chair — Yeditepe University, Health Sciences Faculty, Physiotherapy and Rehabilitation
Locations (1):
- Yeditepe University, Istanbul, Ataşehir, Turkey (Türkiye)